CLINICAL TRIAL: NCT03670615
Title: Exercise Augmenting Cognition tDCS (EXACT): A Pilot Study of a Combined Exercise and Transcranial Direct Current Stimulation Intervention for Cognition
Brief Title: Using Exercise and Electrical Brain Stimulation to Improve Memory in Dementia
Acronym: EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 075-2018
Record Dates: First submitted 2018-08-22; First posted 2018-09-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Alzheimer disease; cognition; transcranial direct current stimulation; exercise; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Motor Activity | interventions — Transcranial Direct Current Stimulation; Exercise; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a randomized, blinded, repeated-session, parallel-design study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The research personnel that will be administering the cognitive assessments will be blinded to treatment allocation. The patients will be blinded to stimulation type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise and tDCS (Experimental): Patients randomized to this group will attend Toronto Rehabilitation Institute - University Health Network (TRI-UHN) for an individualized exercise program and active tDCS intervention.
  Interventions: Other: tDCS; Other: Exercise
- Exercise Education and tDCS (Other): Patients randomized to this group will undergo treatment as usual, receiving routine advice about physical activity and active tDCS intervention.
  Interventions: Other: tDCS; Other: Exercise Education
- Exercise and Sham tDCS (Other): Patients randomized to this group will attend TRI-UHN for an individualized exercise program and sham tDCS intervention.
  Interventions: Other: Exercise; Other: Sham tDCS

INTERVENTIONS:
Other: tDCS — All study participants randomized to tDCS will receive active tDCS.
  Arms: Exercise Education and tDCS; Exercise and tDCS
Other: Exercise — Participants will exercise at TRI according to an individualized exercise prescription.
  Arms: Exercise and Sham tDCS; Exercise and tDCS
Other: Exercise Education — Exercise education/ treatment as usual will include routine advice about physical activity for older adults.
  Other Names: Treatment as usual
  Arms: Exercise Education and tDCS
Other: Sham tDCS — The same procedure for tDCS will be used for the sham condition, except without active current.
  Arms: Exercise and Sham tDCS

SUMMARY:
Mild cognitive impairment and Alzheimer's disease are conditions that involve memory difficulties. Transcranial direct current stimulation is a type of brain stimulation. It may help improve these memory difficulties. However, it works better on active brain areas. This study looks at if combining exercise and applying current to important parts of the brain can help improve memory in people with Mild Cognitive Impairment or Alzheimer's disease.

DETAILED DESCRIPTION:
Objectives: To assess the efficacy of a combined exercise and tDCS treatment for improving cognitive outcomes in mild cognitive impairment and mild Alzheimer's disease.

Study Design: Eligible participants will be randomized to one of three interventions: Exercise and tDCS, Treatment as usual (TAU/exercise education) and tDCS, or Exercise and sham tDCS. Participants randomized to an exercise group will undergo exercise, followed by either sham or active tDCS. Participants randomized to TAU will receive written information in accordance with the Canadian Physical Activity Guidelines for older adults and tDCS for the same duration. Cognition, neuropsychiatric symptoms and blood samples for biomarker analysis will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥50 years of age
* DSM-5 criteria for major or mild neurocognitive disorder due to AD or mixed AD/vascular disease
* Mild severity of impairment (standardized Mini-Mental State Examination (MMSE) score ≥19)
* Read and communicate in English

Exclusion Criteria:

* Change in cognitive enhancing medications (ChEIs and/or memantine) less than 3 months prior to study screen
* Change in anticonvulsants or psychotropic medications less than 1 month prior to study screen
* Currently taking benzodiazepines
* Presence of metal implants that would preclude safe use of tDCS (e.g. pace-maker)
* Significant neurological condition (e.g. epilepsy, Parkinson's disease, multiple sclerosis)
* Current psychiatric disorders (e.g. schizophrenia, bipolar disorder, depression, psychosis) or current substance use disorder
* Medical contraindications to increasing activity level according to the Canadian Society of Exercise Physiology Questionnaire

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Change in cognition: The Word Recognition Task from the Alzheimer's Disease Assessment Scale Cog (ADAS-Cog) | Change over 2 weeks (Baseline to Endpoint)
  Assess recognition memory. Words incorrectly recognized will be tallied. Word Recognition scores range from 0 to 12. Higher scores represent a worse outcome.

SECONDARY OUTCOMES:
Change in cognition: n-back reaction time | Change over 2 weeks (Baseline to Endpoint)
  A measure of working memory. Reaction times in milliseconds will be recorded. Higher values represent a worse outcome.
Change in cognition: The Word Recall Task from the Alzheimer's Disease Assessment Scale-Cog (ADAS-Cog) | Change over 2 weeks (Baseline to Endpoint)
  Assesses recall memory. Number of words not recalled will be tallied. Word recall scores range from 0 to 10. Higher scores represent a worse outcome.
Change in global cognitive function: The Montreal Cognitive Assessment (MoCA) Total Scores | Change over 2 weeks Baseline to Endpoint
  A brief measure of global cognition that includes assessments of orientation, short-term total memory, executive function, language abilities, attention and visuospatial ability. MoCA scores range from 0 to 30. Higher scores represent a better outcome.
Change in neuropsychiatric symptoms: The Neuropsychiatric Inventory (NPI) | Change over 2 weeks (Baseline to Endpoint)
  A widely used assessment of behavior disturbances in dementia including: apathy, agitation, delusions, hallucinations, depression, euphoria, aberrant motor behavior, irritability, disinhibition, anxiety, sleeping, and eating. Frequency and severity of each symptom is measured using subscales. Frequency and severity are judged using a 4-point scale (ranging from 1-4) and 3-point scale (ranging from 1-3) respectively. A 6-point scale for each symptom is used to evaluate caregiver distress (ranging from 0-5). Higher values represent a worse outcome.

OTHER OUTCOMES:
Changes in concentration of blood biomarkers of brain plasticity | Change over 2 weeks (Baseline to Endpoint)
  Biomarkers associated with exercise, tDCS outcomes, angiogenesis and neurogenesis will be obtained from blood work and analyzed using enzyme linked immunosorbent assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Liu CS, Herrmann N, Song BX, Ba J, Gallagher D, Oh PI, Marzolini S, Rajji TK, Charles J, Papneja P, Rapoport MJ, Andreazza AC, Vieira D, Kiss A, Lanctot KL. Exercise priming with transcranial direct current stimulation: a study protocol for a randomized, parallel-design, sham-controlled trial in mild cognitive impairment and Alzheimer's disease. BMC Geriatr. 2021 Dec 4;21(1):677. doi: 10.1186/s12877-021-02636-6. PMID 34863115